CLINICAL TRIAL: NCT01261169
Title: Mycophenolate Sodium (Myfortic®) in the Treatment of Corticosteroid-refractory Autoimmune Uveitis:Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Yih-Shiou Hwang, Yih-Shiou Hwang
Other Study IDs: CERL080ATW06T
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Uveitis
Keywords: Mycophenolate sodium (Myfortic®); Corticosteroid-refractory autoimmune Uveitis
MeSH Terms: conditions — Uveitis | interventions — Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myfortic
  Interventions: Drug: Myfortic

INTERVENTIONS:
Drug: Myfortic — Myfortic in uveitis

SUMMARY:
This study is designed to explore the use of Myfortic® in patients with steroid-refractory uveitis. The aim of the study will be to show the therapeutic effect of Myfortic® in managing uveitis patients.

DETAILED DESCRIPTION:
This study is a single arm prospective evaluation in which patients with uveitis are treated with Myfortic® in a dose of 360 mg bid for six months. From day 0, Myfortic will be combined with 1 mg/kg prednisone. Prednisone will be tapered from week 1 based on the clinical findings of the ophthalmologist.

There will be no other stratification of patients. After the screening, patients will be treated with Myfortic® for 6 months. Patients will be seen at month 1, 3, and 6. Thereafter patients will be followed up at month 12. Efficacy and safety assessments will be performed at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years of age with corticosteroid-refractory uveitis due to one of the inflammatory conditions listed below:

   1. Ocular sarcoidosis: a granulomatous uveitis with posterior inflammation in a patient in which sarcoidosis has been established by means of a biopsy, cytology, or a positive scan.
   2. Intermediate uveitis: patients with clinical features as defined by the IUSG23. However, it is important that the patient has no evidence of a systemic infection such as Lyme Borreliosis and that there is no history of neurological symptoms likely to be associated with multiple sclerosis. All patients with intermediate uveitis should have a negative MRI with gadolinium contrast, prior to being enrolled.
   3. Behçet's syndrome: the international classification criteria of the International Society for Behçet's Disease (ISBD) will be used to define these patients.
   4. Idiopathic Retinal Vasculitis where systemic or infectious causes have been eliminated. In particular patients will not have evidence of Wegener's granulomatosis, SLE, PAN, polymyositis, dermatomyositis or other systemic vasculitic disorders. Patients must also lack evidence for a systemic infection, and have been adequately screened. For the purpose of this study, Eale's disease will be excluded from the idiopathic retinal vasculitis group. However, both non-occlusive and occlusive types of retinal vasculitis can be included in the study.
   5. Vogt-Koyanagi-Harada disease (VKH) as defined according to the international Workgroup definition of VKH.
   6. Sympathetic ophthalmia: a granulomatous uveitis involving the choroid and retina, characterized by multiple white-yellow lesions often in the periphery, which can coalesce particularly in the circumpapillary region. It is associated with trauma or multiple prior surgeries.
   7. Idiopathic panuveitis: all non-infectious panuveititides that can not be related to the diseases mentioned above.
   8. Corticosteroid-refractory uveitis patient is defined as the patient who receive steroid treatment and cannot lower the dosage of steroid to less than 10mg per day in 3 months due to the clinical condition.
2. Disease that is 5 years or less in duration, with a significant flare in the past 24 months requiring intensification of anti-inflammatory therapy (predsinolone). A significant flare is defined as a drop of 2 lines of vision on an ETDRS chart or equivalent, or increase in vitreous flare by 2 grades.
3. Visual acuity of 0.1 or better in at least one eye.
4. Men and women of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicidal cream, or surgical sterilization) for the duration of the study and should continue such precautions for 6 weeks after receiving the last administration.
5. The screening laboratory test results must meet the following criteria:

   1. Hemoglobin ≥ 10.5 g/dL
   2. WBC ≥ 3.0 x 103/μL
   3. Neutrophils ≥ 1.5 x 103/μL
   4. Platelets ≥ 1 x 103/μL
   5. SGOT (AST) and alkaline phosphatase levels must be within 3 times the upper limit of normal range for the laboratory conducting the test (3xULN).
   6. Creatinine clearance > 25 ml/min
6. Must have a normal chest radiograph within 3 months prior to first therapy with no evidence of malignancy, infection or TB.
7. Patient must be able to adhere to the study visit schedule and other protocol requirements.
8. The patient must be capable of giving informed consent and the consent must be obtained prior to any screening procedures.

Exclusion Criteria:

1. Inability to visualize the fundus due to corneal or lenticular opacities.
2. Patients requiring ocular surgery within the initial 3 months of treatment, or who have had surgery in the prior 3 months.
3. Women who are pregnant, nursing, or planning pregnancy within 6 months after screening (i.e., approximately 6 weeks following last treatment).
4. Use of any investigational drug within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
5. Recent history of systemic immunosuppressive therapy, other than steroids for ocular disease within 2 months.
6. Creatinine clearance of < 25ml/min or serum creatinine level higher than 1.5 mg/dl
7. Patients with known hypersensitivity to prednisone, Myfortic® or drugs with similar chemical structures.
8. Patients with any clinically significant infection.
9. Documented HIV infection.
10. Patients with active TB or evidence of latent TB.
11. Patients with positive Lues serology and or significant Lues infection.
12. Patients with opportunistic infections, including but not limited to evidence of active cytomegalovirus, active Pneumocystis carinii, Aspergillosis, Histoplasmosis or atypical mycobacterium infection, etc, within the previous 6 months.
13. Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic,hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
14. Presence of a transplanted organ (with the exception of a corneal transplant 3 months prior to screening).
15. Malignancy within the past 5 years (except for treated squamous or basal cell carcinoma of the skin without evidence of recurrence).
16. History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infra-clavicular, epitrochlear, or periaortic areas), or splenomegaly.
17. Known recent substance abuse (drugs or alcohol).
18. Poor tolerability of venipuncture or lack of adequate venous access for required blood sampling during the study period.
19. Recent live vaccinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 40 patients with uveitis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hwang Yih Shiou, MD, Principal Investigator — CGMH
Locations (1):
- CGMH, Taoyuan, Taiwan, Taiwan